CLINICAL TRIAL: NCT01979133
Title: A Proof of Concept Study of Icariin for Bipolar Disorder and Co-Occurring Substance Use Disorders
Brief Title: Study of Icariin for Bipolar Disorder and Co-Occurring Substance Use Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sherwood Brown, E. Sherwood Brown, M.D., Ph.D., Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 082013-042
Record Dates: First submitted 2013-10-25; First posted 2013-11-08 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder; Substance Use Disorder
MeSH Terms: conditions — Bipolar Disorder; Substance-Related Disorders | interventions — icariin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- icariin (Experimental): Icariin will be given 100 mg/day. A dose titration from 100 mg/day to 200 mg/day will be allowed at week 3 for participants with less than a 30% reduction in HAMD and/or still using cocaine or alcohol or have a positive urine drug screen. An additional dose titration to 300 mg/day will be allowed at week 6 for participants with less than a 50% reduction in HAMD scores and/or still using cocaine or alcohol or have a positive urine drug screen.
  Interventions: Drug: Icariin

INTERVENTIONS:
Drug: Icariin — Participants will receive 20% icariin (100 mg/day) in a commercially available over-the-counter Horny Goat Weed supplement. A dose titration from 100 mg/day to 200 mg/day will be allowed at week 3 participants with less than a 30% reduction in HAMD and/or still using cocaine or alcohol or have a positive urine drug screen. An additional dose titration to 300 mg/day will be allowed at week 6 for participants with less than a 50% reduction in HAMD scores and/or still using cocaine or alcohol or have a positive urine drug screen.
  Other Names: Epimedium, Horny Goat Weed, Yin Yang Huo

SUMMARY:
This study is being done to see if icariin will help with depression in patients with bipolar disorder and alcohol or cocaine use disorders. The pills used in this study contain 20% icariin.

DETAILED DESCRIPTION:
Ten adults with current bipolar disorder (BPD) and current cocaine or alcohol use disorders, based on a structured clinical interview (SCID), and a baseline Hamilton Rating Scale for Depression (HAMD) score of ≥ 15, will be recruited through a patient database of a recently completed study of bipolar disorder patients with cocaine dependence. Informed consent will be obtained. The clinician version of the structured Clinical Interview for DSM-IV (SCID) is a brief structured interview for major Axis I disorders in DSM-IV including major depressive disorder, dysthymic disorder, bipolar disorders, psychotic disorders, anxiety disorders, eating disorders, and alcohol and substance abuse/dependence. This will be given at baseline to confirm bipolar disorder diagnosis. Blood draws and a physical examination by a physician will be performed at baseline to general physical health. Participants will return to receive icariin (100 mg/day)once their general health and diagnosis are confirmed.

Participants will be assessed at baseline and weekly with the HAMD and a urine drug screen, for 8 consecutive weeks after initiating intervention (icariin). A dose titration from 100 mg/day to 200 mg/day will be allowed at week 3 for participants with less than a 30% reduction in HAMD and/or still using cocaine or alcohol or have a positive urine drug screen. An additional dose titration to 300 mg/day will be allowed at week 6 for participants with less than a 50% reduction in HAMD scores and/or still using cocaine or alcohol or have a positive urine drug screen.

Pill counts will be conducted, and a list of current medications and doses will be obtained at each visit. Participants will be compensated and receive bus passes at each appointment. Participants will be evaluated by both the research assistant (RA) and principal investigator (PI) at each follow-up appointment.

The HAM-D will be the primary outcome measure. Other cognitive assessments will be performed at these same visits as well.

ELIGIBILITY:
Inclusion Criteria:

* Current BPD I, II or NOS and cocaine or alcohol use disorder with HAMD score of ≥ 15
* Cocaine or alcohol use with 5 days of initiating study drug
* Men and women
* Age 18-70 years

Exclusion Criteria:

* Psychotic features
* Non-English speakers
* Treatment resistant depression defined as failure of a trial of antidepressants (≥ 4 weeks at a therapeutic dose) in current episode
* Major medical condition including heart, lung, liver or renal disease, cancer, neurological or immunological conditions
* Vulnerable populations including prisoners, cognitively impaired individuals, and pregnant or nursing women
* Prior side effects or allergic reactions to icariin-containing preparations
* Change in psychotropic medications within 14 days of study entry
* Current suicidal ideation (plan and intent), a suicide attempt within the past 12 months or history of > 1 lifetime suicide attempt

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edson S Brown, M.D., Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Icariin
Started | 10
Completed | 7
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Icariin
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Rating Scale of Depression (HAMD) From Baseline to Week 8 (Exit)
Description: HAMD is an observer-rated measure of depressive symptomatology:
  1. 17 questions (answers for individual questions range between 0-3 and 0-4). Total score range: 0-52. No subscales for this measure.
  2. 0 - no depression; 52 - very severe depression (lower score corresponds to a better outcome).
  3. Total score is obtained by summing questions 1-17.
Time Frame: Baseline vs. Week 8 (Exit)
Population: The total enrollment goal was 10. One participant dropped out during the baseline II visit, thus week 8 score was not obtained for that participant and the change from baseline to week 8 could not be collected. Thus, the analysis includes 9 participants instead of proposed 10.
Measure: Mean (Standard Deviation); unit: HAMD scale units
Groups:
- Baseline: Baseline HAMD Score
- Week 8: Week 8 HAMD Score
Arm/Group | Baseline | Week 8
Number analyzed (Participants) | 9 | 9
HAMD scale units | 17.5 (5.2) | 9 (7.4)
Statistical Analysis 1: Comparison: Baseline vs Week 8; Test type: Superiority or Other; p = .012, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Hamilton Rating Scale of Anxiety From Baseline to Week 8 (Exit)
Description: HAMA is a 14-item observer rated measure of anxiety symptomatology:
  1. 14 items in a scale, no subscales. Individual items are score 0 (no anxiety) to 4 (very severe anxiety).
  2. Total scores range from 0-56.
  3. Total scores represent more severe anxiety. Lower scores represent a better outcome.
Time Frame: Baseline vs. Week 8 (Exit)
Population: The planned enrollment was 10 participants. One participant dropped out during Baseline II visit, thus researchers were unable to assess change from baseline to week 8 in this participant. As a results, the overall number of participants analyzed was 9.
Measure: Mean (Standard Deviation); unit: HAMA units on a scale
Groups:
- Baseline: Baseline HAMA Score
- Week 8: Week 8 HAMA Score
Arm/Group | Baseline | Week 8
Number analyzed (Participants) | 9 | 9
HAMA units on a scale | 15.2 (6.4) | 4.6 (6.3)
Statistical Analysis 1: Comparison: Baseline vs Week 8; Test type: Superiority or Other; p = .005, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in Quick Inventory of Depressive Symptomatology (QIDS) Score From Baseline to Week 8
Description: The QIDS is a 16-item self-report measure of depressive symptomatology:
  1. 16 items rated on a scale from 0-3. No subscales for this instrument.
  2. Total score range is 0-27, where higher score represents higher levels of depression. Lower scores associated with better outcomes.
  3. Total score is obtained using the following formula: highest score on items 1-4 + item 5 + highest score on items 6-9 + item 10+item 11+item12+item13+item14+highest score on items 15-16
Time Frame: Baseline vs. Week 8 (Exit)
Population: The planned enrollment was 10 participants. One participant dropped out during Baseline II visit, thus researchers were unable to assess change from baseline to week 8 in this participant. As a result, the overall number of participants included in the analysis was 9.
Measure: Mean (Standard Deviation); unit: QIDS units on a scale
Groups:
- Baseline: Baseline QIDS Score
- Week 8: Week 8 QIDS Score
Arm/Group | Baseline | Week 8
Number analyzed (Participants) | 9 | 9
QIDS units on a scale | 11.8 (5.9) | 5.7 (4.5)
Statistical Analysis 1: Comparison: Baseline vs Week 8; Test type: Superiority or Other; p = .017, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Change in Number of Standard Drinks of Alcohol Per Week Baseline vs. Week 8 (Exit)
Description: 1. Participants are asked to identify the number of alcoholic drinks they consumed on each day within the last 7 days from the day of visit (not including the day of visit). Participants are asked to provide alcohol name and the amount of alcohol they consumed. These values are then converted to standard drinks using a standard drinks calculator.
  2. The minimum number of drinks per week is 0. There is no maximum number of drinks per week, as the maximum number is unique to each participant.
  3. The general convention for standard drinks used in this study is as follows (oz per one standard drink):
     * beer: 12 fl oz (5% ABV)
     * wine: 5 fl oz (10-12% ABV or 18-20% ABV for fortified wine)
     * hard liquor: 1.5 fl oz (40% ABV)
Time Frame: Baseline vs. Week 8 (Exit)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Drinks per week
Groups:
- Baseline: Baseline Mean Standard Drinks Per Week
- Week 8: Week 8 Mean Standard Drinks Per Week
Arm/Group | Baseline | Week 8
Number analyzed (Participants) | 9 | 9
Drinks per week | 38.8 (45.9) | 10.3 (8.2)
Statistical Analysis 1: Comparison: Baseline vs Week 8; Test type: Superiority or Other; p = .038, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Change in Number of Heavy Drinking Days From Baseline to Week 8 (Exit)
Description: 1. Heavy drinking day is defined as 5 standard drinks per day for men, and 4 standard drinks per day for women.
  2. Minimum score is 0 (no drinks); maximum score is unique to each individual participant. Lower score represents a better outcome.
  3. Average number of heavy drinking days per week is calculated by asking participants to identify the number of drinks they had on each day during the past 7 days (not including the day of visit).
  4. See outcome measure description for "standard drinks per week" for standard drinks convention.
Time Frame: Baseline vs. Week 8 (Exit)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days Per Week
Groups:
- Baseline: Baseline Heavy Drinking Days Per Week
- Week 8: Week 8 Heavy Drinking Days Per Week
Arm/Group | Baseline | Week 8
Number analyzed (Participants) | 9 | 9
Days Per Week | 3.2 (2.0) | 1.2 (1.2)
Statistical Analysis 1: Comparison: Baseline vs Week 8; Test type: Superiority or Other; p = .034, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Change in Days of Alcohol Use From Baseline to Week 8 (Exit)
Description: 1. Total score range is 0-7 (no days of alcohol use - 7 days of alcohol use). The lower score represents better outcome.
  2. Participants are asked to identify days on which they used alcohol in the past week (not including the day of visit).
Time Frame: Baseline vs. Week 8 (Exit)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Days Per Week
Groups:
- Baseline: Baseline Days of alcohol use per week
- Week 8: Week 8 Days of alcohol use per week
Arm/Group | Baseline | Week 8
Number analyzed (Participants) | 9 | 9
Days Per Week | 4.1 (2.4) | 3.3 (1.0)
Statistical Analysis 1: Comparison: Baseline vs Week 8; Test type: Superiority or Other; p = .231, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Change in Young Mania Rating Scale (YMRS) From Baseline to Week 8 (Exit)
Description: The YMRS is an 11-item observer-rated measure of mania symptomatology:
  1. 7 individual items are scored between 0-4.
  2. 4 individual items are scored between 0-8.
  3. Total score range is 0-60, with no subscales. Higher score is indicative of more manic symptoms. Lower score represents better outcomes.
  4. Total score is obtained by adding items on the scale together.
Time Frame: Baseline vs. Week 8 (Exit)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: YMRS units on a scale
Groups:
- Baseline: Baseline YMRS Score
- Week 8: Week 8 YMRS Score
Arm/Group | Baseline | Week 8
Number analyzed (Participants) | 9 | 9
YMRS units on a scale | 8.8 (7.0) | 3.3 (3.5)
Statistical Analysis 1: Comparison: Baseline vs Week 8; Test type: Superiority or Other; p = .066, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Icariin
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No